CLINICAL TRIAL: NCT00337038
Title: Endothelial Function as a Marker for Blood Pressure Control Among Hypertensive Diabetic Patients
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Soroka University Medical Center (Other)
Responsible Party: Principal Investigator, Valentin Yurkevich, Dr Yurkevich, Soroka University Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: sor431706ctil
Record Dates: First submitted 2006-06-14; First posted 2006-06-15 (Estimated); Last update posted 2012-06-22 (Estimated); Status verified 2012-06

CONDITIONS: Hypertension; Diabetes Mellitus Type 2
MeSH Terms: conditions — Hypertension; Diabetes Mellitus, Type 2 | interventions — Acetylcysteine

INTERVENTIONS:
Drug: N-acetylcystein(drug) — p.O t.Siran 200mg x1 during one weak
  Other Names: siran

SUMMARY:
Our aim is to examine the influence of blood pressure and glycemic control together with N-acetylcystein utilization on the endothelia function of hypertensive diabetic patient.The study population will include 50 diabetic patient with uncontrolled hypertention that will be recruited from the Hypertension Clinic of Soroka University Medical Center.

ELIGIBILITY:
Inclusion Criteria:

* Diabetic patients with uncontrolled hypertension that will be recruited from the Hypertension Clinic of Soroka University Medical Center

Exclusion Criteria:

* Pregnancy,secondary hypertention,malignancy or other serious illness

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2006-06; Primary Completion 2010-07 (Actual); Study Completion 2010-07 (Actual)

PRIMARY OUTCOMES:
endothelial function | half of year

SECONDARY OUTCOMES:
blood pressure and glycemic control | half of year

CONTACTS AND LOCATIONS:
Overall Officials: Ester Paran, MD, Principal Investigator — Hypertension Clinic of Soroka University Medical Center; Ester Paran, MD, Principal Investigator — Soroka University Medical Center